CLINICAL TRIAL: NCT03538756
Title: walk2Wellness: Long-term Use Effects of Walkasins® Wearable Sensory Prosthesis on Gait Function, Balance-Confidence, and Social Participation
Brief Title: walk2Wellness: Long-term Effects of Walkasins® Wearable Sensory Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxFunction Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CIP 0002 & CIP 0003
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Sensory Peripheral Neuropathy; Balance; Distorted; Sensation Disorders
Keywords: Balance; Peripheral Neuropathy; Neuropathy
MeSH Terms: conditions — Sensation Disorders; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized only during the baseline visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Baseline Group A--Walkasins On Then Off (Experimental): Subjects will first wear Walkasins and receive vibrotactile feedback that reflects real changes in center of pressure sway. Following a one-hour rest period, they will be retested with Walkasins turned off.
  After the baseline visit, subjects will take the devices home for long-term use and return for periodic follow-up visits
  Interventions: Device: Walkasins
- Baseline Group B--Walkasins Off Then On (Experimental): Subjects will first wear Walkasins turned off and not receive any vibrotactile feedback. Following a one-hour rest period, they will be retested with Walkasins turned on.
  After the baseline visit, subjects will take the devices home for long-term use and return for periodic follow-up visits.
  Interventions: Device: Walkasins
- Single Arm Long-Term Follow-up (Experimental): During the baseline visit, participants were randomized to two groups that applied to the first visit only. After the baseline visit, community-dwelling participants received Walkasins to wear over the next 52 weeks. They returned for follow-up visits at weeks 2, 6, 10, 26, and 52, during which they repeated the functional measures while wearing their Walkasins and responded to the questionnaires. Between weeks 10 and 26 and 26 and 52, they were contacted periodically to remind them of study requirements and to collect follow-up information regarding health changes, adverse events, pain scores, device usage, and device functioning.
  Note: Due to COVID-19 disruptions, some participants were not able to return for all in-person follow-up visits. They completed the patient-reported outcome measures via telephone visits.
  Interventions: Device: Walkasins

INTERVENTIONS:
Device: Walkasins — Walkasins® consist of two parts for each leg: the Haptic Module (leg unit) and the Receptor Sole (foot pad). The Haptic Module wraps around the lower leg of the user and contains electronics for reading Receptor Sole pressure signals, a microprocessor, and four vibrating motors that provide gentle tactile sensory cues to the front, back, medial, and lateral surfaces of the user's leg. These cues reflect real-time foot pressure information at a location above the ankle where skin sensation is still present.

SUMMARY:
The purpose of this study is to investigate the long-term effects of Walkasins® use on clinical and subject-reported outcomes of balance and gait function, quality of life, physical activity/participation, pain, and medication use in persons with peripheral neuropathy who experience balance problems.

DETAILED DESCRIPTION:
The main objectives of this single-arm study are to show a long-term (10 weeks), sustained improvement in Functional Gait Assessment (FGA) score >4 following Walkasins use as compared to participants' initial baseline assessments and to examine a potential relationship between initial baseline assessment data and long-term outcomes. The previous finding of a short-term FGA change >4 during Walkasins use (NCT02115633) justifies a pre-post study design to investigate the long-term effects of Walkasins use. Although the primary timeframe for the primary endpoint is 10 weeks, participants will return for follow-up visits at 26 weeks and 52 weeks of Walkasins use.

The investigators also intend to extend their observations of the short-term effects of Walkasins by replicating the randomized cross-over design of a previous short-term study. (The randomized cross-over replication will occur only during the baseline visit. The long-term study consists of a single arm.) This study may help to further refine the prescription criteria for Walkasins and determine whether or not the presence of a short-term response is indicative of long-term improvements.

A subset of 10 participants at the Harvard Medical School site will be enrolled in a pilot study to investigate possible structural and functional changes in cortical areas of the brain related to somatosensory connectivity using magnetic resonance imaging (MRI). Structural as well as functional MRI scans will be acquired at baseline and after 26 weeks of daily Walkasins use. An exploratory analysis of MRI data will be performed and related to functional clinical outcomes associated with Walkasins use over the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-90 years, male or female
* Formal diagnosis of sensory peripheral neuropathy prior to participating in the study
* Self-reported balance problems
* Ability for transfers or ambulation on level surfaces at fixed cadence as assessed by the physical therapist during the FGA
* FGA <23, the cut-off score for high fall-risk
* Ability to understand and provide informed consent
* Foot size that allows Walkasins® to function appropriately
* Must be able to complete all functional outcome measures without the use of an assistive device

Exclusion Criteria:

* Inability to perceive vibration from Walkasins leg unit
* Use of ankle-foot orthosis for ambulation that prevents donning of Walkasins
* Acute thrombophlebitis including deep vein thrombosis
* Untreated lymphedema
* Untreated lesion of any kind, swelling, infection, inflamed area of skin or eruptions on the lower leg near product use
* Untreated fractures in the foot and ankle
* Severe peripheral vascular disease
* Musculoskeletal or other neurological conditions that prohibit use of Walkasins as determined by clinician
* Weighs more than 300 pounds
* Plans to begin balance physical therapy (PT) during the first ten weeks of the clinical trial (Ongoing or previous balance PT is not an exclusionary criterion.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Oddsson, PhD, Study Director — RxFunction Inc.
Locations (5):
- United States (5):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Marcus Institute for Aging Research, Harvard Medical School, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Fairview Health Services, Saint Paul, Minnesota
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oddsson LIE, Bisson T, Cohen HS, Iloputaife I, Jacobs L, Kung D, Lipsitz LA, Manor B, McCracken P, Rumsey Y, Wrisley DM, Koehler-McNicholas SR. Extended effects of a wearable sensory prosthesis on gait, balance function and falls after 26 weeks of use in persons with peripheral neuropathy and high fall risk-The walk2Wellness trial. Front Aging Neurosci. 2022 Sep 20;14:931048. doi: 10.3389/fnagi.2022.931048. eCollection 2022. PMID 36204554
- [Derived] Oddsson LIE, Bisson T, Cohen HS, Jacobs L, Khoshnoodi M, Kung D, Lipsitz LA, Manor B, McCracken P, Rumsey Y, Wrisley DM, Koehler-McNicholas SR. The Effects of a Wearable Sensory Prosthesis on Gait and Balance Function After 10 Weeks of Use in Persons With Peripheral Neuropathy and High Fall Risk - The walk2Wellness Trial. Front Aging Neurosci. 2020 Nov 9;12:592751. doi: 10.3389/fnagi.2020.592751. eCollection 2020. PMID 33240077
- See also: Sponsor Website — http://rxfunction.com/index.php/contact/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at five sites through various methods, including physician referral and recruitment posters. The first participant was enrolled on October 22, 2018, and the last participant was enrolled in April 2021.
Pre-assignment Details: Sixty-nine participants met the eligibility criteria and received Walkasins, the study device, to be worn on both feet for the duration of their participation. Primary reasons for exclusion were participants' inability to feel the Walkasins stimuli, participants' need of an assistive device to complete the functional assessments, or FGA scores 23 or higher, indicating only limited gait impairments.
Groups:
- Baseline Cross-over Group A--Walkasins ON Then OFF: Subjects will first wear Walkasins and receive vibrotactile feedback that reflects real changes in center of pressure sway. Following a one-hour rest period, they will be retested with Walkasins turned off.
  After the baseline visit, subjects will take the devices home for long-term use and return for periodic follow-up visits.
- Baseline Cross-over Group B--Walkasins OFF Then ON: Subjects will first wear Walkasins turned off and not receive any vibrotactile feedback. Following a one-hour rest period, they will be retested with Walkasins turned on.
  After the baseline visit, subjects will take the devices home for long-term use and return for periodic follow-up visits.
- Single-Arm Long-Term Follow-up (Walkasins ON): The randomized cross-over group assignments applied only to the baseline visit. After the baseline visit, participants received Walkasins to wear over the next 52 weeks. They returned for follow-up visits at weeks 2, 6, 10, 26, and 52. Between weeks 10 and 26 and 26 and 52, they were contacted periodically to remind them of study requirements and to collect follow-up information regarding health changes, adverse events, pain scores, and device usage and functioning.
Period: Baseline Cross-over
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Started | 36 | 33 | 0
Completed | 36 | 33 | 0
Not Completed | 0 | 0 | 0
Period: Long-Term Follow-up
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Started | 0 | 0 | 69
Completed (Week 52 Follow-up Visit) | 0 | 0 | 36
Not Completed | 0 | 0 | 33
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — COVID-19 Disruptions at Sites | 0 | 0 | 13
Not completed — Device Dissatisfaction | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Single-Arm Long-Term Use: After the baseline visit, participants will receive Walkasins to wear over the next 52 weeks. They will return for follow-up visits at weeks 2, 6, 10, 26, and 52. Between weeks 10 and 26 and 26 and 52, they will be contacted periodically to remind them of study requirements and to collect follow-up information regarding health changes, adverse events, pain scores, device usage, and device functioning.
Arm/Group | Single-Arm Long-Term Use
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 69
Weight (kg) [Mean (Standard Deviation); unit: Kilograms] | 89.7 (18.2)

OUTCOME MEASURES:

1. Primary Outcome: Functional Gait Assessment
Description: The Functional Gait Assessment (FGA) is a 10-item scale that measures postural stability while individuals perform walking tasks that are scored from 0 to 3 (3 = normal, 2 = mild impairment, 1 = moderate impairment, 0 = severe impairment). Scores range from a minimum of 0 to a maximum of 30. Higher scores indicate better postural stability. (Participants scoring 23 or higher on the baseline FGA were not included in this study because their peripheral neuropathy was not yet affecting their gait/balance significantly.)
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: Because of study disruptions due to COVID-19, some participants were unable to attend in-person visits; others withdrew from the study for various reasons. The data reported at Weeks 2, 6, 10, 26, and 52 (the protocol-specified assessment times) reflect only the active participants who completed the outcome measure at the specified timepoint. (The protocol stated that no imputation methods would be used to infer missing values of any outcome measures.)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 14.8 (4.1) | 14.8 (4.1) | 14.8 (4.1)
  Baseline Crossover--Walkasins ON: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins ON | 17.0 (4.5) | 18.2 (3.8) |
  Baseline Crossover--Walkasins OFF: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins OFF | 17.14 (4.5) | 16.3 (3.9) |
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 17.9 (4.7)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 18.2 (4.4)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 19.2 (5)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 19.1 (4)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 20.7 (5.3)

2. Secondary Outcome: 10-Meter Walk Test
Description: Gait speed (10-meter walk, timing the middle 6 meters) is assessed under two conditions: Participants are instructed (1) to walk at normal speed and (2) to walk as fast as they can. Higher numbers indicate faster speeds (i.e., more meters per second).
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters/Second
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
Meters/Second
  Baseline Normal Gait Speed | 0.90 (0.29) | 0.85 (0.19) | 0.88 (0.25)
  Baseline Crossover--Walkasins ON: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins ON | 0.92 (0.28) | 0.91 (0.19) |
  Baseline Crossover--Walkasins OFF: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins OFF | 0.95 (0.29) | 0.90 (0.17) |
  Week 2 Normal Gait Speed: number analyzed (Participants) | 0 | 0 | 60
  Week 2 Normal Gait Speed |  |  | 0.94 (0.28)
  Week 6 Normal Gait Speed: number analyzed (Participants) | 0 | 0 | 55
  Week 6 Normal Gait Speed |  |  | 0.95 (0.27)
  Week 10 Normal Gait Speed: number analyzed (Participants) | 0 | 0 | 51
  Week 10 Normal Gait Speed |  |  | 0.97 (0.26)
  Week 26 Normal Gait Speed: number analyzed (Participants) | 0 | 0 | 44
  Week 26 Normal Gait Speed |  |  | 0.97 (0.28)
  Week 52 Normal Gait Speed: number analyzed (Participants) | 0 | 0 | 36
  Week 52 Normal Gait Speed |  |  | 1.02 (0.30)

3. Secondary Outcome: Timed Up and Go Test (TUG)
Description: The Timed Up and Go Test is part of the Centers for Disease Control (CDC)-recommended STEADI test protocol for balance function. From a seated position in a standard armchair, the participant is asked to stand up from the chair, walk to a line on the floor 10 feet away at normal pace, turn, walk back to the chair at normal pace, and sit down again. The tester records the time taken from the command "Go" until the subject sits down again. Lower times indicate better/faster performance.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
Seconds
  Baseline | 13.9 (6.2) | 13.5 (4.5) | 13.7 (5.5)
  Baseline Crossover--Walkasins ON: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins ON | 13.7 (5.2) | 12.8 (3.9) |
  Baseline Crossover--Walkasins OFF: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins OFF | 13.2 (5.8) | 12.7 (3.7) |
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 12.8 (4.2)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 12.4 (4.2)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 12.1 (3.6)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 12.3 (3.4)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 12.2 (3.7)

4. Secondary Outcome: Four-Stage Balance Test
Description: The 4-Stage Balance Test is part of the Centers for Disease Control's recommended test protocol for balance function. It includes four gradually more challenging postures the subject is exposed to: (1) Stand with feet side by side. (2) Stand with feet in semi-tandem stance. (3) Stand with feet in tandem stance. (4) Stand on one leg. Participants pass each level if they can hold the stance for 10 seconds and then move on to the next stance. If they cannot hold the stance, the test ends. Higher times indicate better balance than lower times.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
Seconds
  Baseline | 24.2 (6.9) | 26.5 (8.0) | 25.3 (7.5)
  Baseline Crossover--Walkasins ON: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins ON | 25.4 (7.5) | 26.6 (6.4) |
  Baseline Crossover--Walkasins OFF: number analyzed (Participants) | 36 | 33 | 0
  Baseline Crossover--Walkasins OFF | 26.0 (6.9) | 27.7 (6.6) |
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 27.1 (8.0)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 27.4 (7.4)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 27.3 (6.9)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 28.4 (5.6)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 31.1 (6.8)

5. Secondary Outcome: Activities-specific Balance Confidence (ABC) Scale
Description: Powell and Myers (1995) developed the Activities-specific Balance Confidence (ABC) Scale to detect levels of balance confidence in elderly persons. The ABC scale is a one-page questionnaire that asks questions about balance confidence when performing 16 different tasks. The items are rated on a scale of 0 to 100; a score of 0 indicates no confidence and a score of 100 indicates complete confidence when performing the task. The overall score is calculated by adding the individual items then dividing by the total number of items (16). The higher the score, the greater the person's balance confidence; thus, higher scores indicate that subjects are more confident of their balance.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: IBecause of study disruptions due to COVID-19, some participants were unable to attend in-person visits; others withdrew from the study for various reasons. The data reported at Weeks 2, 6, 10, 26, and 52 (the protocol-specified assessment times) reflect only the active participants who completed the outcome measure at the specified timepoint. (The protocol stated that no imputation methods would be used to infer missing values of any outcome measures.)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline Crossover | 58.2 (17.3) | 61.2 (16.2) | 59.6 (16.7)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 62.5 (15.2)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 62.3 (16.9)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 63.6 (14.8)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 62.1 (16.5)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 65.2 (16.7)

6. Secondary Outcome: Vestibular Activities of Daily Living Scale (VADL)
Description: The Vestibular Activities of Daily Living Scale (VADL) is a self-reported questionnaire that was developed to assess self-perceived disability in individuals with vestibular impairment. It evaluates the effects of vertigo and balance disorders on independence in 28 activities of daily living. Participants selected a number ranging from 1 = "Independent" to 10 = "Too Difficult, No Longer Perform." The scores on the 28 activities were averaged. The higher the score (up to 10), the greater is the person's self-perceived disability (i.e., the person feels less independence in activities of daily living). Lower averages of the 28 items indicate greater independence in activities of daily living (e.g., a healthy adult's VADL score most likely would be between 1.0 and 2.0).
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 3.97 (1.13) | 3.82 (1.15) | 3.89 (1.14)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 3.49 (1.1)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 3.66 (1.09)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 3.78 (1.03)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 3.66 (1.22)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 3.62 (1.12)

7. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a nine-question tool for assessing depression and emotional well-being. Participants rate nine areas on a 0 to 3 scale in response to the question, "Over the last 2 weeks, how often have you been bothered by any of the following problems?" The rating scale is as follows: 0 = "Not at All," 1 = "Several Days," 2 = "More Than Half the Days," and 3 = "Nearly Every Day." A PHQ-9 total score of 0-4 points indicates "normal" or minimal depression. Scores between 5-9 points indicate mild depression; 10-14 points, moderate depression; 15-19 points, moderately severe depression; and 20 or more points, severe depression. (The minimum score on the PHQ-9 is 0; the maximum score is 27.) In short, lower scores indicate less depression.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 5.19 (4.63) | 4.30 (3.53) | 4.77 (4.13)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 3.97 (3.96)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 4.12 (4.16)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 4.18 (4.62)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 4.19 (4.03)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 4.83 (4.95)

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 6b
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 6b measures the self-reported consequences of pain on relevant aspects of a person's life over the past 7 days and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. PROMIS measures are scored on the T-score metric (mean = 50, standard deviation = 10). Higher scores (i.e., those greater than 50, the mean) indicate that the participants perceive their pain as interfering in their daily lives more than average; lower scores (i.e., those less than 50, the mean) indicate that the participants perceive their pain as interfering less than average in their daily lives, which would be considered a better outcome.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
T-score
  Baseline | 52.6 (8.3) | 50.1 (8.7) | 51.4 (8.5)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 51.7 (7.8)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 51.1 (8.9)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 52.2 (8.5)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 51.2 (8.5)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 52.8 (9.1)

9. Secondary Outcome: PROMIS Pain Intensity Form 1a
Description: The PROMIS Pain Intensity Form 1a instrument asks participants to rate the intensity of their pain on average over the previous 7 days. It is universal rather than disease specific. The higher the score on a scale of 0 ("no pain") to 10 ("worst pain imaginable), the more intense is the person's perception of pain; lower scores indicate less intense perception of pain, a better outcome.
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 3.2 (2.6) | 2.4 (2.0) | 2.8 (2.3)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 2.6 (2.1)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 2.8 (2.5)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 2.7 (2.4)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 2.7 (2.1)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 3.2 (2.9)

10. Secondary Outcome: PROMIS Ability to Participate Short Form 8a
Description: The PROMIS Ability to Participate in Social Roles and Activities assesses the participants' perceived ability to perform their usual social roles and activities. PROMIS measures are scored on the T-score metric (mean = 50, standard deviation = 10). A higher score (i.e., greater than 50, the mean) indicates participants perceive they have a better ability to participate in their roles and activities (i.e., a better outcome).
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 48.8 (7.7) | 50.7 (8.7) | 49.7 (8.2)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 51.1 (7.5)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 50.9 (7.3)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 51.1 (7.9)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 52.0 (8.1)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 48.7 (7.9)

11. Secondary Outcome: PROMIS Satisfaction With Participation in Social Roles Short Form 8a
Description: The PROMIS Satisfaction with Social Roles and Activities items assess satisfaction with performing one's usual social roles and activities (e.g., "I am satisfied with my ability to participate in family activities"). PROMIS measures are scored on the T-score metric (mean = 50, standard deviation = 10). A higher score (i.e., those greater than 50, the mean) indicates the respondents' greater satisfaction in regard to their ability to participate in their roles and activities (i.e., a better outcome).
Time Frame: Baseline, Week 2, Week 6, Week 10 (Primary Endpoint), Week 26, and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 36 | 33 | 69
score on a scale
  Baseline | 47.7 (6.3) | 49.9 (8.1) | 48.7 (7.3)
  Week 2: number analyzed (Participants) | 0 | 0 | 60
  Week 2 |  |  | 49.2 (7.5)
  Week 6: number analyzed (Participants) | 0 | 0 | 55
  Week 6 |  |  | 50.1 (7.9)
  Week 10: number analyzed (Participants) | 0 | 0 | 51
  Week 10 |  |  | 50.4 (8.4)
  Week 26: number analyzed (Participants) | 0 | 0 | 44
  Week 26 |  |  | 51.0 (8.3)
  Week 52: number analyzed (Participants) | 0 | 0 | 36
  Week 52 |  |  | 49.4 (8.5)

12. Secondary Outcome: Falls
Description: Subjects were asked about the number of times they have fallen in the past 6 and 12 months and whether they incurred an injury from falling. (For this study, the researchers used the World Health Organization's definition of a fall: "an event which results in a person coming to rest inadvertently on the ground or floor or other lower level.") These data were compared to falls during their participation in the trial as tracked with a calendar and reported as adverse events. Falls data were monitored as overall number of falls and fallers pre-and post-study participation as well as the number of falls/1000 patient days. A lower number indicates fewer falls over 26 weeks (6 months).
Time Frame: Baseline and 26 Weeks
Population: Data on falls were collected and analyzed for 44 participants who completed at least 26 weeks of the study. (At baseline subjects reported the number of falls they had experienced in the six months prior to their participation in the trial.)
Measure: Number; unit: Number of Participant Falls
Groups:
- Baseline Cross-over Group A--Walkasins ON Then OFF; Baseline Cross-over Group B--Walkasins OFF Then ON; Single-Arm Long-Term Follow-up (Walkasins ON): The randomized cross-over group assignments applied only to the baseline visit. After the baseline visit, participants received Walkasins to wear over the next 52 weeks. They returned for follow-up visits at weeks 2, 6, 10, 26, and 52. Between weeks 10 and 26 and 26 and 52, they were contacted periodically to remind them of study requirements and to collect follow-up information regarding health changes, adverse events, pain scores, and device usage and functioning.
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
Number analyzed (Participants) | 0 | 0 | 44
Number of Participant Falls
  Pre-Study/Baseline |  |  | 53
  Week 26 |  |  | 39

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the period of each subject's participation, a maximum of 52 weeks per participant. (The average duration of subjects' participation in the study was 271 days.)
Description: The randomized cross-over assignments applied only to the baseline visit. Adverse events were not collected or analyzed by the randomized groups; they were collected for all participants in the single arm long-term portion of this study.
Groups:
- Single-Arm Long-Term Follow-up (Walkasins ON): During the baseline visit, participants were randomized to two groups that applied to the first visit only. After the baseline visit, all the participants received Walkasins to wear over the next 52 weeks (single arm). They returned for follow-up visits at weeks 2, 6, 10, 26, and 52. Between weeks 10 and 26 and 26 and 52, they were contacted periodically to remind them of study requirements and to collect follow-up information regarding health changes, adverse events, pain scores, device usage, and device functioning.
Arm/Group | Baseline Cross-over Group A--Walkasins ON Then OFF | Baseline Cross-over Group B--Walkasins OFF Then ON | Single-Arm Long-Term Follow-up (Walkasins ON)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 1/69
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 10/69
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 24/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Cross-over Group A--Walkasins ON Then OFF (N=0) | Baseline Cross-over Group B--Walkasins OFF Then ON (N=0) | Single-Arm Long-Term Follow-up (Walkasins ON) (N=69)
Hospitalizations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (5) — Hospitalizations were for atrial flutter and atrial fibrillation; they were unrelated to device use.
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (3) — Hospitalizations were for pneumonia/respiratory problems; they were unrelated to device use.
Hospitalizations (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) — Hospitalizations were for hip fractures; they were unrelated to device use.
Hospitalization (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) — Hospitalization was for critical anemia; it was unrelated to device use.
Hospitalization (Cardiac disorders) | 0 | 0 | 1 (1) — Hospitalization was for severe hypotension; it was unrelated to device use.
Hospitalization (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) — Hospitalization was for low magnesium; it was unrelated to device use.
Hospitalization (Psychiatric disorders) | 0 | 0 | 1 (1) — Hospitalization was for mental health; it was unrelated to device use.
Hospitalization (Surgical and medical procedures) | 0 | 0 | 1 (1) — Hospitalization was for a surgical procedure; it was unrelated to device use.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Cross-over Group A--Walkasins ON Then OFF (N=0) | Baseline Cross-over Group B--Walkasins OFF Then ON (N=0) | Single-Arm Long-Term Follow-up (Walkasins ON) (N=69)
Falls with Minor Injuries (General disorders) | 0 | 0 | 24 (48) — This study collected information on falls, per the World Health Organization (WHO) definition. Minor injuries included scrapes and bruises. Many participants suffered from comorbidities and used medications that may have impacted their balance.
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 (4)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 (7)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 (12) — Skin irritation includes blisters, cracked skin, rashes, etc. on participants' feet or lower legs.

LIMITATIONS AND CAVEATS:
The main limitations of this trial were the following: (1) It was not blinded, and it lacked a control group and a placebo treatment. (2) We enrolled a greater percentage of males than females. (3) Lockdowns at the study sites due to COVID-19 caused significant disruptions to data collection for the functional measures. Some participants also indicated that COVID-19 impacted their daily activities, which, in turn, affected the amount of time they used the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the principal results from any single center experience within the study can occur following the preparation and publication of the multicenter results. (This restriction no longer applies since the multicenter results have been published.)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT03538756/Prot_SAP_000.pdf